CLINICAL TRIAL: NCT01143740
Title: An Exploratory Biomarker Study of RO5045337 in Patients With Liposarcomas Prior to Debulking Surgery
Brief Title: A Study of RO5045337 in Patients With Liposarcomas Prior to Debulking Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP22890; 2009-015522-10
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: RO5045337

INTERVENTIONS:
Drug: RO5045337 — orally day 1-10 each 28-day cycle, 3 cycles

SUMMARY:
This open-label study will evaluate efficacy, safety and tolerability of RO5045337 in patients with liposarcoma who are eligible for debulking surgery. Prior to surgery, patients will receive 2-3 cycles of RO5045337, orally for 10 days followed by 18 days of rest per cycle. Anticipated time on study treatment is 3 months. Patients with an incomplete resection may be treated for an additional 3 cycles with RO5045337.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=18 years of age
* well differentiated and/or dedifferentiated liposarcoma eligible for tumor debulking surgery
* willing to undergo tumor biopsies before, during and after treatment
* ECOG performance status 0-1

Exclusion Criteria:

* previous chemotherapy and/or radiation for liposarcoma; previous debulking surgery is acceptable
* patients receiving any other agent or therapy to treat their malignancy
* patients requiring anticoagulant therapy and/or anti-platelet therapy
* pre-existing gastrointestinal disorders which may interfere with absorption of drugs
* history of seizure disorders or unstable CNS metastases
* clinically significant cardiovascular disease
* history of long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Biomarker evidence of MDM2 and p53 pathway alterations (histologic, molecular and imaging analyses) | from baseline to week 12

SECONDARY OUTCOMES:
Safety and tolerability: Adverse events, laboratory parameters, ECG | up to approximately 4 months after study start
Tumor response according to RECIST criteria assessed by CT or MRI | from baseline to week 7
Correlation pharmacokinetics (AUC, Cmax, tmax, t1/2, CL/V, V/F) - pharmacodynamics/biomarkers | multiple sampling weeks 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- France (4):
  - Bordeaux
  - Lille
  - Lyon
  - Villejuif